CLINICAL TRIAL: NCT04561271
Title: Feasability of Foot Reflexology to Alleviate Anxiety in Palliative Care Unit : a Pilot Randomised Double Blind Study
Brief Title: Feasability of Foot Reflexology to Alleviate Anxiety in Palliative Care Unit (RPASP)
Acronym: RPASP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RBHP 2020 GUASTELLA; 2020-A01880-39 (Other: ANSM)
Record Dates: First submitted 2020-09-08; First posted 2020-09-23 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: End Stage Disease
Keywords: Palliative care; Foot reflexology; Anxiety; Acceptability; Feasability
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: 2 arms, one called "foot reflexology" who receive one session, the second called "toucher massage".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- foot reflexology (Experimental): patients will receive one session of foot reflexology with a nurse who received a specific formation. The session lasts 15 to 20 minutes, patients seated, half seated or in supine position. The technique consists in stimulating reflex zones of foot, each zone corresponding to a specific organ. Almond oil will be used. The session is accompanied by relaxing music
  Interventions: Other: foot reflexology
- toucher massage (Sham Comparator): patients will receive one session of toucher massage with a nurse (this technique is taught during the formation of every nurse in palliative care units). The session lasts 15 to 20 minutes, patients seated, half seated or in supine position. It consists in a simple massage and effleurage, with fluid and progressive movements. Almond oil will be used. The session is accompanied by relaxing music.
  Interventions: Other: toucher massage

INTERVENTIONS:
Other: foot reflexology — Patients will receive one session of foot reflexology with a nurse who received a specific formation. The session lasts 15 to 20 minutes, patients seated, half seated or in supine position. A neutral oil will be used. The technique associates specific movements of foot reflexology. The session is accompanied by relaxing music.
  Arms: foot reflexology
Other: toucher massage — one session of toucher massage with a nurse (this technique is taught during the formation of every nurse in palliative care units). The session lasts 15 to 20 minutes, patients seated, half seated or in supine position. It consists in a simple massage and effleurage, with fluid and progressive movements. Almond oil will be used. The session is accompanied by relaxing music.
  Arms: toucher massage

SUMMARY:
The primary purpose of the study is to know if foot reflexology can be accepted by patients hospitalized in palliative unit care (assessed by the number of patient who accept to participate), and if it is feasible (assessed by the realization of one session in normal condition : duration of 15-20 min, in supine position/seated or half-seated position).The investigators make the hypothesis that patients will accept to receive foot reflexology, and maybe feel less anxious after one session.

DETAILED DESCRIPTION:
The patients will receive an informative content about the study and will have 24 hours of reflexion. If they accept to participate to the study, they will be randomised in one of the two groups : foot reflexology or "toucher massage" (for those randomised in the "toucher massage" group, a session of foot reflexology will be proposed in a second time). The investigators will assess the level of anxiety, the quality of the sleep and the pain using the ESAS scale, before and after the session. 24 hours after the session, they will be interviewed about what they felt with the session. The investigators will also have a look on the anxiolytic and antagic medication they consume before and after the session.

ELIGIBILITY:
Inclusion Criteria:

* Adult able to give consent, man or woman, hospitalized in palliative care unit, with vigilance criteria from +1 to -3 on the Richmond scale.
* Affiliated to Social Security

Exclusion Criteria:

* Painfull bone metastasis on the feet
* foot amputation
* foot bedsore
* peripheral distal neuropathy, trouble of foot sensibility
* agonic or pre agonic state
* Patients under juridical protection
* Refusal to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
acceptability of foot reflexology in palliative care unit | day 0
  the acceptability will be assessed by the number of patient who accept to participate to the study
feasibility of foot reflexology in palliative care unit | day 0
  The feasibility will be assessed by the conditions of realization of one session : for the study, the normal conditions will be : duration (15-20 min) and possibility for the patient to remain in the good position (supine position/seated or half-seated position).

SECONDARY OUTCOMES:
Effects of foot reflexology on anxiety | Before the session (day 0) and 24 hours after
  investigator will assess the anxiety, using the Edmonton Symptom Assessment System (ESAS scale), before and after the session. This scale permits the patient to choose a number from 0 to 10, 0 corresponding to the lowest level of anxiety, and 10 corresponding to the highest level of anxiety
Effects of foot reflexology on pain | Before the session (day 0) and 24 hours after
  investigators will assess the pain using the Edmonton Symptom Assessment System (ESAS scale), before and after the session. This scale permits the patient to choose a number from 0 to 10, 0 corresponding to the lowest level of pain, and 10 corresponding to the highest level of pain
Effects of foot reflexology on sleep quality | Before the session (day 0) and 24 hours after
  investigators will assess the sleep quality using the Edmonton Symptom Assessment System (ESAS scale), before and after the session. This scale permits the patient to choose a number from 0 to 10, 0 corresponding to the lowest level of tiredness, and 10 corresponding to the highest level of tiredness.
Effects of foot reflexology on anxiolytic intake | Before the session (day 0) and 24 hours after
  investigators will write down the anxiolytic intake before the session, and until 24 hours after the session, using redcap software. There will be a "yes/no" question for "benzodiazepine" and "neuroleptic". If "yes" is chosen, there will be a free text box to be more specific
Effects of foot reflexology on pain killers intake | Before the session (day 0) and 24 hours after
  investigators will write down the pain killer intake before the session, and until 24 hours after the session, using redcap software. There will be a "yes/no" question for "paracetamol", "weak opioids", "strong opioids" and "co-analgesics". If "yes" is chosen, there will be a free text box to be more specific.
patients' experience | day 1
  24 hours after the session, investigators will collect patients' experience and feeling about the session they undergone. Key words and verbatims will be reported on a free text box with redcap

CONTACTS AND LOCATIONS:
Overall Officials: Virginie Guastella, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France